CLINICAL TRIAL: NCT04331574
Title: Phase IV Observational Study to Associate Hypertension and Hypertensinon Treatment to COVID19
Brief Title: Renin-Angiotensin System Inhibitors and COVID-19
Acronym: SARS-RAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Societa Italiana dell'Ipertensione Arteriosa (Other)
Responsible Party: Sponsor
Other Study IDs: SARS-RAS
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Hypertension; Cardiovascular Diseases
Keywords: risk factors; SARS; ACE Inibitors; ARB
MeSH Terms: conditions — COVID-19; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid-19 patients: Patients with certified diagnosis of COVID-19 recruited in Italian hospitals

SUMMARY:
Multicentric non-profit observational study, in patients with COVID-19 hospitalized in Italy, conducted through a pseudonymised survey.

DETAILED DESCRIPTION:
The recent SARS-CoV-2 Coronavirus pandemic and subsequent spread of the disease called COVID-19 brought back to the discussion a topic already highlighted during the SARS-CoV-4 crown-related SARS epidemic of 2002. In particular, the angiotensin converting enzyme 2 (ACE2) has been identified as a functional receptor for coronaviruses, therefore including SARS-CoV-2. ACE2 is strongly expressed in the heart and lungs. SARS-CoV-2 mainly invades alveolar epithelial cells, resulting in respiratory symptoms. These symptoms could be made more severe in the presence of increased expression of ACE2. ACE2 levels can be increased by the use of renin-angiotensin system inhibitors (RAS). This therapeutic class is particularly widespread, as it represents the most important pharmacological protection for widespread diseases such as high blood pressure, heart failure and ischemic heart disease. It is therefore possible to hypothesize that pharmacological treatment with RAS inhibitors may be associated with a more severe symptomatology and clinic than COVID-19.

However, several observations from studies on SARSCoV, which are most likely also relevant for SARS-CoV-2 seem to suggest otherwise. Indeed, it has been shown that the binding of coronavirus to ACE2 leads to downregulation of ACE2, which in turn causes an ACE / ACE2 imbalance excessive production of angiotensin by the related ACE enzyme. Angiotensin II receptor 1 (AT1R) stimulated by angiotensin causes an increase in pulmonary vascular permeability, thereby mediating an increase in lung damage. Therefore, according to this hypothesis, the upregulation of ACE2, caused by the chronic intake of AT1R and ACE Inhibitors, could be protective through two mechanisms: the first, that of blocking in the AT1 receptor; second, increasing ACE2 levels decreases ACE production of angiotensin and increases ACE2 production of angiotensin 1-7.

The quickest approach to evaluating these two opposing hypotheses is to analyze the medical records of COVID-19 patients to determine whether patients on RAS antagonist therapy have a different disease outcome than patients without the above therapy.

This research aims to verify whether the chronic intake of RAS inhibitors modifies the prevalence and severity of the clinical manifestation of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Patients affected by COVID19 referring to italian outpatient clinics or hospitals

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients enrolled in infectious disease and resuscitation centers in Italy or in home isolation and health surveillance
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of COVID-19 patients enrolled that use ACE inhibitors and/or Angiotensin Receptor Blockers (ARB) as antihypertensive agents | 3 months
  Using anamnestic data collected from the health record of the hospital or of the general practitioner, we will count the number of COVID-19 patients enrolled that were treated with ACE Inhibitors or ARB.
Numbers of COVID-19 patients enrolled with no symptoms, with moderate symptoms or with severe symptoms of pneumoni based on the WHO specification for ARDS that also used ACE inhibitors and/or Angiotensin Receptor Blockers (ARB) as antihypertensive agents | 3 months
  This study want to observe whether the assumption of antihypertensive ACE inhibitors or ARB increases the severity of the clinical manifestation of COVID19

SECONDARY OUTCOMES:
Number and type of anthropometric and clinical parameters that associate with COVID19 and COVID-19 severity | 3 months
  Collecting selected data from the health record and hospital charts of the patients we will assess whether among the recorded parameters there are any that can predict COVID19 prevalence and severity

CONTACTS AND LOCATIONS:
Overall Officials: Guido Iaccarino, MD, Study Chair — Federico II University; Guido Grassi, MD, Study Director — Inversity of Milan, BICOCCA; MariaLorenza Muiesan, MD, Principal Investigator — Università degli Studi di Brescia; Claudio Borghi, MD, Principal Investigator — University of Bologna; Claudio Ferri, MD, Principal Investigator — University of L'Aquila; MASSIMO VOLPE, MD, Principal Investigator — Univerity of Rome "La Sapienza"; Leonardo Sechi, Principal Investigator — University of Udine
Locations (1):
- Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iaccarino G, Grassi G, Borghi C, Grassi D, Mancusi C, Muiesan ML, Salvetti M, Volpe M, Ferri C. Preexisting Oral Anticoagulant Therapy Ameliorates Prognosis in Hospitalized COVID-19 Patients. Front Cardiovasc Med. 2021 May 13;8:633878. doi: 10.3389/fcvm.2021.633878. eCollection 2021. PMID 34055928
- [Derived] Iaccarino G, Grassi G, Borghi C, Carugo S, Fallo F, Ferri C, Giannattasio C, Grassi D, Letizia C, Mancusi C, Minuz P, Perlini S, Pucci G, Rizzoni D, Salvetti M, Sarzani R, Sechi L, Veglio F, Volpe M, Muiesan ML; SARS-RAS Investigators. Gender differences in predictors of intensive care units admission among COVID-19 patients: The results of the SARS-RAS study of the Italian Society of Hypertension. PLoS One. 2020 Oct 6;15(10):e0237297. doi: 10.1371/journal.pone.0237297. eCollection 2020. PMID 33022004
- [Derived] Iaccarino G, Grassi G, Borghi C, Ferri C, Salvetti M, Volpe M; SARS-RAS Investigators. Age and Multimorbidity Predict Death Among COVID-19 Patients: Results of the SARS-RAS Study of the Italian Society of Hypertension. Hypertension. 2020 Aug;76(2):366-372. doi: 10.1161/HYPERTENSIONAHA.120.15324. Epub 2020 Jun 22. PMID 32564693
- See also: Related Info — https://siia.it/notizie-siia/inibitori-del-sistema-renina-angiotensina-e-sars-cov-2-lindagine-della-siia/